CLINICAL TRIAL: NCT00002470
Title: A Phase II Study of Protracted Infusional 5-Fluorouracil Plus Alpha Interferon for Advanced Metastatic Carcinoid
Brief Title: Fluorouracil Plus Interferon Alfa in Treating Patients With Advanced Metastatic Carcinoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mid-Atlantic Oncology Program (Other)
Collaborators: Cancer Biotherapy Research Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MAOP-5190; CDR0000076667 (Registry Identifier: PDQ (Physician Data Query)); NBSG-9010; NCI-V90-0197
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2003-12

CONDITIONS: Gastrointestinal Carcinoid Tumor; Lung Cancer
Keywords: metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; pulmonary carcinoid tumor
MeSH Terms: conditions — Lung Neoplasms | interventions — Interferon-alpha; Fluorouracil

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of the cancer cells. Combining interferon alfa with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of fluorouracil plus interferon alfa in treating patients who have advanced metastatic carcinoid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate and duration of remission in patients with advanced metastatic carcinoid tumors treated with fluorouracil and interferon alfa-2b.
* Determine the symptomatic response in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.
* Determine the survival characteristics of patients treated with this regimen.

OUTLINE: Patients receive fluorouracil IV continuously for 10 weeks and interferon alfa subcutaneously 3 times a week for 12 weeks. Treatment continues every 12 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and at weeks 1, 7, and 11 of each course.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven carcinoid tumor with radiologically confirmed metastatic disease
* Recurrence after surgery or radiotherapy allowed
* Must meet at least 1 of the following conditions:

  * Symptomatic carcinoid syndrome not controlled
  * Other systemic symptoms (e.g., weight loss, anorexia)
  * 24 hour urinary 5-hydroxyindole acetic acid (5-HIAA) 100 mg or greater
  * Bone metastases
  * Carcinoid heart disease
  * Carcinoid asthma
* Measurable disease or 24-hour urinary 5-HIAA 50 mg or greater required
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 3.0 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* See Disease Characteristics

Pulmonary:

* See Disease Characteristics

Other:

* No concurrent infection (no fever for at least 3 days prior to treatment unless fever due to tumor)
* No significant medical or psychiatric illness that would preclude study or informed consent
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or curatively treated stage I carcinoma of the cervix
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior interferon therapy

Chemotherapy:

* No other concurrent chemotherapy

Endocrine therapy:

* Prior endocrine therapy allowed
* Concurrent octreotide allowed

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Prior surgery allowed

Other:

* No prior fluorinated pyrimidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1990-09; Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Ahlgren, MD, Study Chair — George Washington University; Robert K. Oldham, MD, Study Chair — Cancer Therapeutics, Incorporated
Locations (1):
- George Washington University Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Ahlgren JD, Leming PD, Gullo JJ, et al.: Protracted infusional 5-FU (PIF) + alpha2b-interferon (alpha-IFN) in metastatic carcinoid: updated experience with Mid-Atlantic Oncology Program (MAOP) study 5190. [Abstract] Proceedings of the American Society of Clinical Oncology 14: A-552, 219, 1995.
- [Result] Ahlgren JD, Leming PD, Fryer D, et al.: Protracted infusional 5-FU (PIF) + alpha2b-interferon (alpha-IFN): a well tolerated regimen for palliation of advanced carcinoid: a Mid-Atlantic Oncology Program (MAOP) study. [Abstract] Proceedings of the American Society of Clinical Oncology 12: A-661, 218, 1993.